CLINICAL TRIAL: NCT01444430
Title: A 26 Week, Randomized, Double-blind, Parallel-group, Active Controlled, Multicenter, Multinational Safety Study Evaluating the Risk of Serious Asthma-related Events During Treatment With Symbicort®, a Fixed Combination of Inhaled Corticosteroid (ICS) (Budesonide) and a Long Acting β2-agonist (LABA) (Formoterol) as Compared to Treatment With ICS (Budesonide) Alone in Adult and Adolescent (≥12 Years of Age) Patients With Asthma
Brief Title: A 6 Month Safety Study Comparing Symbicort With Inhaled Corticosteroid Only in Asthmatic Adults and Adolescents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D5896C00027; 2011-002790-28 (EudraCT Number)
Record Dates: First submitted 2011-09-23; First posted 2011-09-30 (Estimated); Results first posted 2016-12-15 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-11

CONDITIONS: Asthma
Keywords: Symbicort pMDI; Asthma; safety; budesonide
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental): Symbicort
  Interventions: Drug: Symbicort pMDI
- 2 (Active Comparator): budesonide
  Interventions: Drug: budesonide pMDI

INTERVENTIONS:
Drug: Symbicort pMDI — Patients were randomized to Symbicort and assigned to one of the following treatments (based upon ACQ at baseline and prior asthma therapy): Symbicort pMDI 80/4.5 μg x 2 actuations bid (morning and evening) or Symbicort pMDI 160/4.5 μg x 2 actuations bid (morning and evening), for oral inhalation.
  Arms: 1
Drug: budesonide pMDI — Patients were randomized to budesonide and assigned to one of the following treatments (based upon ACQ at baseline and prior asthma therapy): budesonide pMDI 80 μg x 2 actuations bid (morning and evening) or budesonide pMDI 160 μg x 2 actuations bid (morning and evening), for oral inhalation.
  Arms: 2

SUMMARY:
The purpose of the study is to evaluate the safety of Symbicort compared to inhaled corticosteroid alone during 6 months in adult and adolescent patients with asthma

DETAILED DESCRIPTION:
A 26 week, randomized, double-blind, parallel-group, active controlled, multicenter, multinational safety study evaluating the risk of serious asthma-related events during treatment with Symbicort®, a fixed combination of inhaled corticosteroid (ICS) (budesonide) and a long acting β2-agonist (LABA) (formoterol) as compared to treatment with ICS (budesonide) alone in adult and adolescent (≥12 years of age) patients with asthma.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed informed consent/ paediatric assent (if applicable) prior to any study specific procedures including medication withdrawal
* Male or Female, ≥12 years of age
* Documented clinical diagnosis of asthma for at least 1 year prior to Visit 2
* Patient must have history of at least 1 asthma exacerbation including one of the following:

  * requiring treatment with systemic corticosteroids
  * an asthma-related hospitalization between 4 weeks and 12 months prior to randomization
* Current Asthma Therapy: Patients must be appropriately using one of the treatments for asthma listed in the protocol combined with achieving certain results when recording an Asthma Control Questionnaire

Exclusion Criteria:

* Patient has a history of life-threatening asthma. Defined for this protocol as an asthma episode that required intubation and/or was associated with hypercapnea requiring non-invasive ventilatory support.
* Patient has required treatment with systemic corticosteroids (tablets, suspensions or injectable) for any reason within 4 weeks prior to Visit 2
* Patient has an ongoing exacerbation, defined as a worsening of asthma that requires treatment with systemic corticosteroids (tablets, suspension, or injectable)
* An asthma exacerbation within 4 weeks of randomization or more than 4 separate exacerbations in the 12 months preceding randomization or more than 2 hospitalizations for treatment of asthma in the 12 months preceding randomization
* Patient has a respiratory infection or other viral/bacterial illness, or is recovering from such an illness at the time of Visit 2 that, in the investigator's opinion, will interfere with the patient's lung function
* Patient must not meet unstable asthma severity criteria as listed in the protocol
* Peak expiratory flow must not be below 50% o predicted normal
* Pregnancy, breast-feeding or planned pregnancy during the study

Ages: 12 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12460 (Actual)
Dates: Start 2011-12; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carin Jorup, Study Director — AstraZeneca Pepparedsleden 1, 431 83 Mölndal
Locations (340):
- United States (160):
  - Research Site, Birmingham, Alabama
  - Research Site, Huntsville, Alabama
  - Research Site, Anchorage, Alaska
  - Research Site, Gilbert, Arizona
  - Research Site, Glendale, Arizona
  - Research Site, Mesa, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Fort Smith, Arkansas
  - Research Site, Little Rock, Arkansas
  - Research Site, Alhambra, California
  - Research Site, Anaheim, California
  - Research Site, Arvin, California
  - Research Site, Bellflower, California
  - Research Site, Buena Park, California
  - Research Site, Costa Mesa, California
  - Research Site, Encinitas, California
  - Research Site, Escondido, California
  - Research Site, Fountain Valley, California
  - Research Site, Glendale, California
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Newport Beach, California
  - Research Site, Northridge, California
  - Research Site, Palmdale, California
  - Research Site, Pasadena, California
  - Research Site, Poway, California
  - Research Site, Riverside, California
  - Research Site, Roseville, California
  - Research Site, San Diego, California
  - Research Site, San Jose, California
  - Research Site, Santa Ana, California
  - Research Site, Stockton, California
  - Research Site, Tustin, California
  - Research Site, Walnut Creek, California
  - Research Site, Denver, Colorado
  - Research Site, Thornton, Colorado
  - Research Site, Norwalk, Connecticut
  - Research Site, Waterbury, Connecticut
  - Research Site, Altamonte Springs, Florida
  - Research Site, Clearwater, Florida
  - Research Site, DeLand, Florida
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Fort Myers, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Kissimmee, Florida
  - Research Site, Leesburg, Florida
  - Research Site, Lehigh Acres, Florida
  - Research Site, Lynn Haven, Florida
  - Research Site, Miami, Florida
  - Research Site, Miami Beach, Florida
  - Research Site, Ocoee, Florida
  - Research Site, Opa-locka, Florida
  - Research Site, Orlando, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Royal Palm Beach, Florida
  - Research Site, Tampa, Florida
  - Research Site, Calhoun, Georgia
  - Research Site, Conyers, Georgia
  - Research Site, Decatur, Georgia
  - Research Site, Gainesville, Georgia
  - Research Site, Savannah, Georgia
  - Research Site, Hayden Lake, Idaho
  - Research Site, Meridan, Idaho
  - Research Site, Kenilworth, Illinois
  - Research Site, Springfield, Illinois
  - Research Site, Anderson, Indiana
  - Research Site, Evansville, Indiana
  - Research Site, Michigan City, Indiana
  - Research Site, Ames, Iowa
  - Research Site, Council Bluffs, Iowa
  - Research Site, Fort Mitchell, Kentucky
  - Research Site, Lexington, Kentucky
  - Research Site, Owensboro, Kentucky
  - Research Site, Lafayette, Louisiana
  - Research Site, Lake Charles, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Lanham, Maryland
  - Research Site, Watertown, Massachusetts
  - Research Site, Kalamazoo, Michigan
  - Research Site, Madison Hgts, Michigan
  - Research Site, Port Huron, Michigan
  - Research Site, Southfield, Michigan
  - Research Site, Sterling Heights, Michigan
  - Research Site, Ypsilanti, Michigan
  - Research Site, Duluth, Minnesota
  - Research Site, Edina, Minnesota
  - Research Site, Biloxi, Mississippi
  - Research Site, Jackson, Mississippi
  - Research Site, Vicksburg, Mississippi
  - Research Site, Bridgeton, Missouri
  - Research Site, Chesterfield, Missouri
  - Research Site, Kansas City, Missouri
  - Research Site, Springfield, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Bellevue, Nebraska
  - Research Site, Grand Island, Nebraska
  - Research Site, Omaha, Nebraska
  - Research Site, Verona, New Jersey
  - Research Site, Great Neck, New York
  - Research Site, Hopewell Jct, New York
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, Rockville Centre, New York
  - Research Site, The Bronx, New York
  - Research Site, Watertown, New York
  - Research Site, Cary, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Salisbury, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Fargo, North Dakota
  - Research Site, Cincinnati, Ohio
  - Research Site, Miamishburg, Ohio
  - Research Site, Stow, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Bend, Oregon
  - Research Site, Abington, Pennsylvania
  - Research Site, Bryn Mawr, Pennsylvania
  - Research Site, Doylestown, Pennsylvania
  - Research Site, Phoenixville, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Wyomissing, Pennsylvania
  - Research Site, Warwick, Rhode Island
  - Research Site, Charleston, South Carolina
  - Research Site, Greeneville, South Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, Greer, South Carolina
  - Research Site, Old Point Station, South Carolina
  - Research Site, Summerville, South Carolina
  - Research Site, Knoxville, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Baytown, Texas
  - Research Site, Dallas, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Georgetown, Texas
  - Research Site, Houston, Texas
  - Research Site, Killeen, Texas
  - Research Site, McKinney, Texas
  - Research Site, Pharr, Texas
  - Research Site, Plano, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Spring, Texas
  - Research Site, Sugar Land, Texas
  - Research Site, Sugarland, Texas
  - Research Site, Waco, Texas
  - Research Site, Layton, Utah
  - Research Site, South Burlington, Vermont
  - Research Site, Danville, Virginia
  - Research Site, Vienna, Virginia
  - Research Site, Virginia Beach, Virginia
  - Research Site, Seattle, Washington
  - Research Site, Spokane, Washington
  - Research Site, Tacoma, Washington
  - Research Site, La Crosse, Wisconsin
  - Research Site, Milwaukee, Wisconsin
- Argentina (8):
  - Research Site, Buenos Aires
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Córdoba
  - Research Site, Mar del Plata
  - Research Site, Monte Grande
  - Research Site, Quilmes
  - Research Site, Ranelagh
  - Research Site, San Miguel de Tucumán
- Brazil (7):
  - Research Site, Barueri
  - Research Site, Botucatu
  - Research Site, Goiânia
  - Research Site, Juiz de Fora
  - Research Site, Porto Alegre
  - Research Site, Santo André
  - Research Site, São Paulo
- Bulgaria (13):
  - Research Site, Gotse Delchev
  - Research Site, Kozloduy
  - Research Site, Petrich
  - Research Site, Pleven
  - Research Site, Razgrad
  - Research Site, Razlog
  - Research Site, Rousse
  - Research Site, Sandanski
  - Research Site, Sevlievo
  - Research Site, Sofia
  - Research Site, Stara Zagora
  - Research Site, Varna
  - Research Site, Vidin
- Chile (3):
  - Research Site, Quillota
  - Research Site, Santiago
  - Research Site, Viña del Mar
- Colombia (3):
  - Research Site, Bogotá
  - Research Site, Cali
  - Research Site, Manizales
- Czechia (9):
  - Research Site, Beroun
  - Research Site, Břeclav
  - Research Site, Krnov
  - Research Site, Kutná Hora
  - Research Site, Litoměřice
  - Research Site, Ostrava
  - Research Site, Pilsen
  - Research Site, Prague
  - Research Site, Rokycany
- France (3):
  - Research Site, Angers
  - Research Site, Perpignan
  - Research Site, Tiercé
- Germany (4):
  - Research Site, Berlin
  - Research Site, Hamburg
  - Research Site, Leipzig
  - Research Site, Marburg
- India (10):
  - Research Site, Bangalore
  - Research Site, Calicut
  - Research Site, Coimbatore
  - Research Site, Goa
  - Research Site, Hyderabad
  - Research Site, Mangalore
  - Research Site, Mysore
  - Research Site, Nagpur
  - Research Site, New Delhi
  - Research Site, Trivandrum
- Italy (9):
  - Research Site, Benevento
  - Research Site, Bologna
  - Research Site, Catanzaro
  - Research Site, Ferrara
  - Research Site, Genova
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Palermo
  - Research Site, Roma
- Mexico (8):
  - Research Site, Durango
  - Research Site, Guadalajara
  - Research Site, México
  - Research Site, Monterrey
  - Research Site, Morelia
  - Research Site, Querétaro City
  - Research Site, Villahermosa
  - Research Site, Zapopan
- Research Site, Panama City, Panama
- Peru (2):
  - Research Site, Cusco
  - Research Site, Lima
- Philippines (5):
  - Research Site, Iloilo City
  - Research Site, Lipa City
  - Research Site, Manila
  - Research Site, Pasig
  - Research Site, Quezon City
- Poland (14):
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Chęciny
  - Research Site, Gorzów Wlkp
  - Research Site, Karpacz
  - Research Site, Krakow
  - Research Site, Ostrów Wielkopolski
  - Research Site, Skarżysko-Kamienna
  - Research Site, Strzelce Opolskie
  - Research Site, Szczecin
  - Research Site, Tarnów
  - Research Site, Turek
  - Research Site, Urszulin
  - Research Site, Wroclaw
- Puerto Rico (3):
  - Research Site, Caguas
  - Research Site, San Juan
  - Research Site, Toa Baja
- Romania (9):
  - Research Site, Bragadiru
  - Research Site, Brasov
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Constanța
  - Research Site, Craiova
  - Research Site, Deva
  - Research Site, Iași
  - Research Site, Tg. Mures
- Russia (11):
  - Research Site, Kazan'
  - Research Site, Moscow
  - Research Site, Novosibirsk
  - Research Site, Penza
  - Research Site, Saint Petersburg
  - Research Site, Saratov
  - Research Site, StPetersburg
  - Research Site, Vladikavkaz
  - Research Site, Volgograd
  - Research Site, Yaroslavl
  - Research Site, Yekaterinburg
- Slovakia (12):
  - Research Site, Bardejov
  - Research Site, Bratislava
  - Research Site, Dunajská Streda
  - Research Site, Komárno
  - Research Site, Košice
  - Research Site, Liptovský Mikuláš
  - Research Site, Nitra
  - Research Site, Prešov
  - Research Site, Ružomberok
  - Research Site, Skalica
  - Research Site, Zvolen
  - Research Site, Žilina
- South Africa (10):
  - Research Site, Boksburg North
  - Research Site, Breyten
  - Research Site, Cape Town
  - Research Site, Durban
  - Research Site, eMkhomazi
  - Research Site, Johannesburg
  - Research Site, Lenasia
  - Research Site, Lyttleton
  - Research Site, Pretoria
  - Research Site, Verulam
- South Korea (6):
  - Research Site, Ansan-si
  - Research Site, Cheonan-si
  - Research Site, Cheongju-si
  - Research Site, Jinju
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Thailand (5):
  - Research Site, Bangkok
  - Research Site, Hat Yai
  - Research Site, Khon Kaen
  - Research Site, Muang,
  - Research Site, Naimuang
- Ukraine (10):
  - Research Site, Dnipropetrovsk
  - Research Site, Donetsk
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv
  - Research Site, Kiev
  - Research Site, Odesa
  - Research Site, Poltava
  - Research Site, Uzhhorod
  - Research Site, Vinnitsa
  - Research Site, Zaporozye
- United Kingdom (13):
  - Research Site, Bath
  - Research Site, Belfast
  - Research Site, Blackpool
  - Research Site, Canterbury
  - Research Site, Chippenham
  - Research Site, Coventry
  - Research Site, Crawley
  - Research Site, Leicester
  - Research Site, Royal Leamington Spa
  - Research Site, Stockport
  - Research Site, Trowbridge
  - Research Site, Watford
  - Research Site, Westbury
- Vietnam (2):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City

REFERENCES:
- [Derived] Peters SP, Bleecker ER, Canonica GW, Park YB, Ramirez R, Hollis S, Fjallbrant H, Jorup C, Martin UJ. Serious Asthma Events with Budesonide plus Formoterol vs. Budesonide Alone. N Engl J Med. 2016 Sep 1;375(9):850-60. doi: 10.1056/NEJMoa1511190. PMID 27579635
- See also: D5896C00027_Protocol_redacted.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=541&filename=D5896C00027_Protocol_redacted.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study started with an assessment visit where inclusion/exclusion criteria were reviewed and informed consent obtained. Eligible patients were randomized at the next visit. Patients then entered a 26 weeks double-blind treatment period followed by a 1 week follow-up telephone contact. Patients were recruited in 25 countries with 25% in the US.
Pre-assignment Details: Eligible adult and adolescent patients were stratified based upon assessment of ACQ and prior asthma therapy and randomized 1:1 to double-blind Symbicort or budesonide. 12460 patients were enrolled (informed consent received) and 11693 were randomized.
Groups:
- Symbicort: Patients were randomized to Symbicort and assigned to one of the following treatments (based upon ACQ at baseline and prior asthma therapy): Symbicort pMDI 80/4.5 μg x 2 actuations bid (morning and evening) or Symbicort pMDI 160/4.5 μg x 2 actuations bid (morning and evening).
- Budesonide: Patients were randomized to budesonide and assigned to one of the following treatments (based upon ACQ at baseline and prior asthma therapy): budesonide pMDI 80 μg x 2 actuations bid (morning and evening) or budesonide pMDI 160 μg x 2 actuations bid (morning and evening).
Period: Overall Study
Arm/Group | Symbicort | Budesonide
Started | 5846 | 5847
Completed | 5785 | 5766
Not Completed | 61 | 81
Not completed — Withdrawal by Subject | 53 | 72
Not completed — Death | 6 | 8
Not completed — Lost to Follow-up | 2 | 0
Not completed — CRF termination module not completed. | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Symbicort | Budesonide | Total
Number analyzed (Participants) | 5846 | 5847 | 11693
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.4 (17.4) | 43.5 (17.3) | 43.5 (17.3)
Gender [Count of Participants; unit: Participants]
  Female | 3849 | 3820 | 7669
  Male | 1997 | 2027 | 4024
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 4050 | 4003 | 8053
  Black/African American | 396 | 401 | 797
  Asian | 848 | 907 | 1755
  Native Hawaiian/Pacific Islander | 3 | 3 | 6
  American Indian/Alaska Native | 225 | 207 | 432
  Other | 324 | 326 | 650

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing an Event in the Composite Endpoint (Asthma-related Death, Asthma-related Intubation or Asthma-related Hospitalization)
Description: Number of participants experiencing an event in the composite endpoint (asthma-related death, asthma-related intubation or asthma-related hospitalization), using events adjudicated and confirmed by the Joint Adjudication Committee. Cox proportional hazards model with terms for randomized treatment and strata for incoming control/asthma treatment was used to compare Symbicort and budesonide. Hazard ratios and 95% confidence intervals were estimated.
Time Frame: Up to 27 weeks
Population: Full analysis set (FAS) population comprised of all patients randomized to study drug.
Measure: Number; unit: Participants
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 5846 | 5847
Participants | 43 | 40
Statistical Analysis 1: Comparison: Symbicort vs Budesonide; Test type: Non-Inferiority or Equivalence — The upper limit of the 95% CI of the hazard ratio will be used to assess statistical non-inferiority (non-inferiority margin=2); Regression, Cox; Hazard Ratio (HR) = 1.073, 95% CI 2-sided [0.698 to 1.650]

2. Primary Outcome: Number of Participants Experiencing an Event Included in the Definition of Asthma Exacerbation
Description: Number of participants experiencing an event included in the definition of asthma exacerbation. An asthma exacerbation was defined as a deterioration of asthma requiring systemic corticosteroids for at least 3 days or an inpatient hospitalization or emergency room visit due to asthma that required systemic corticosteroids. Cox proportional hazards model with terms for randomized treatment and strata for incoming control/asthma treatment was used to compare Symbicort and budesonide. Hazard ratios and 95% confidence intervals were estimated.
Time Frame: Up to 26 weeks
Population: The On treatment Analysis set comprised of all randomized patients and included data that corresponded to each patient's period of exposure to study drug plus 7 days after the last date of study drug treatment.
Measure: Number; unit: Participants
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 5846 | 5847
Participants | 539 | 633
Statistical Analysis 1: Comparison: Symbicort vs Budesonide; Test type: Superiority or Other; p = 0.002, Regression, Cox; Hazard Ratio (HR) = 0.835, 95% CI 2-sided [0.745 to 0.937]

3. Secondary Outcome: Percent of Days With no Asthma Symptoms
Description: Percent of days with no asthma symptoms during the randomized treatment period. Analysis of variance (ANOVA) model including the fixed factors of treatment and strata by incoming control/asthma treatment was used to compare Symbicort and budesonide.
Time Frame: Daily up to 26 weeks
Population: Full analysis set (FAS) population comprised of all patients randomized to study drug and had at least one entry of diary data after randomization.
Measure: Least Squares Mean (Standard Error); unit: Percentage of days
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 5784 | 5796
Percentage of days | 81.1 (0.4) | 76.8 (0.4)
Statistical Analysis 1: Comparison: Symbicort vs Budesonide; Test type: Superiority or Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 4.4, 95% CI 2-sided [3.3 to 5.4], Standard Error of Mean 0.5

4. Secondary Outcome: Percent of Days With Activity Limitation Due to Asthma
Description: Percent of days with activity limitation due to asthma during the randomized treatment period. Analysis of variance (ANOVA) model including the fixed factors of treatment and strata by incoming control/asthma treatment was used to compare Symbicort and budesonide.
Time Frame: Daily up to 26 weeks
Population: Full analysis set (FAS) population comprised of all patients randomized to study drug. The analysis set comprises of all patients with at least one day with asthma symptoms, i.e. the denominator is the number of days with asthma symptoms.
Measure: Least Squares Mean (Standard Error); unit: Percentage of days
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 4895 | 5045
Percentage of days | 19.7 (0.4) | 19.1 (0.4)
Statistical Analysis 1: Comparison: Symbicort vs Budesonide; Test type: Superiority or Other; p = 0.272, ANOVA; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-0.5 to 1.7], Standard Error of Mean 0.6

5. Secondary Outcome: Mean Number of Puffs of Rescue Medication Per 24 Hours
Description: Mean number of puffs of rescue medication per day (24 hours) during the randomized treatment period. Analysis of variance (ANOVA) model including the fixed factors of treatment and strata by incoming control/asthma treatment was used to compare Symbicort and budesonide.
Time Frame: Daily up to 26 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Inhalations/day
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 5784 | 5796
Inhalations/day | 0.8 (0.0) | 0.9 (0.0)
Statistical Analysis 1: Comparison: Symbicort vs Budesonide; Test type: Superiority or Other; p < 0.001, ANOVA; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.2 to -0.1], Standard Error of Mean 0.0

6. Secondary Outcome: Asthma Control Questionnaire (ACQ6)
Description: The outcome variable for ACQ6 was the difference between the average of values recorded during the treatment period (day 28, day 84 and day 182) and the baseline measure. Analysis of covariance (ANCOVA) model, including the fixed factors of treatment and strata by incoming control/asthma treatment and baseline ACQ6 as covariate was used to compare Symbicort and budesonide.
  The asthma control questionnaire, ACQ6, consists of six questions; all assessed on a 7-point scale from 0 to 6, where 0 represents good control and 6 represents poor control. The overall score is the mean of the responses to each of the six questions.
Time Frame: baseline, day 28, day 84, day 182
Population: Full analysis set (FAS) population comprised of all patients randomized to study drug with at least one post-baseline ACQ6 score.
Measure: Least Squares Mean (Standard Error); unit: ACQ6 overall score change from baseline
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 5701 | 5698
ACQ6 overall score change from baseline | -0.70 (0.01) | -0.62 (0.01)
Statistical Analysis 1: Comparison: Symbicort vs Budesonide; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-0.10 to -0.06], Standard Error of Mean 0.01

7. Secondary Outcome: Percent of Nights With Awakening(s) Due to Asthma
Description: Percent of nights with awakening(s) due to asthma during the randomized treatment period. Analysis of variance (ANOVA) model including the fixed factors of treatment and strata by incoming control/asthma treatment was used to compare Symbicort and budesonide.
Time Frame: Daily up to 26 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Percentage of nights
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 5784 | 5796
Percentage of nights | 4.0 (0.2) | 4.7 (0.2)
Statistical Analysis 1: Comparison: Symbicort vs Budesonide; Test type: Superiority or Other; p = 0.004, ANOVA; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-1.0 to -0.2], Standard Error of Mean 0.2

8. Secondary Outcome: Number of Participants Experiencing Discontinuation of Investigational Product Due to a Protocol Defined Asthma Exacerbation
Description: Number of participants experiencing discontinuation of investigational product due to a protocol defined asthma exacerbation. An asthma exacerbation was defined as a deterioration of asthma requiring systemic corticosteroids for at least 3 days or an inpatient hospitalization or emergency room visit due to asthma that required systemic corticosteroids. Cox proportional hazards model with terms for randomized treatment and strata for incoming control/asthma treatment was used to compare Symbicort and budesonide. Hazard ratios and 95% confidence intervals were estimated.
Time Frame: Up to 26 weeks
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 5846 | 5847
Participants | 53 | 71
Statistical Analysis 1: Comparison: Symbicort vs Budesonide; Test type: Superiority or Other; p = 0.095, Regression, Cox; Hazard Ratio (HR) = 0.739, 95% CI 2-sided [0.518 to 1.055]

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and discontinuation of treatment with investigational product due to adverse event (DAEs) were recorded from the time of informed consent through the treatment period and including the follow-up period, up to 27 weeks.
Description: AEs were not collected unless they lead to discontinuation or qualified as an SAE.
Arm/Group | Symbicort | Budesonide
Serious Adverse Events (participants affected / at risk) | 125/5846 | 123/5847
Other Adverse Events (participants affected / at risk) | 0/5846 | 0/5847
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Symbicort (N=5846) | Budesonide (N=5847)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Angina pectoris (Cardiac disorders) | 3 (3) | 1 (1)
Angina unstable (Cardiac disorders) | 2 (2) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 3 (3)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery insufficiency (Cardiac disorders) | 0 (0) | 1 (1)
Hypertensive heart disease (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 3 (3)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Erosive oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 2 (2)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intussusception (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 1 (1)
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1)
Device dislocation (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 2 (2)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biliary dyskinesia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Allergic granulomatous angiitis (Immune system disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Anaphylactic shock (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Bronchitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0)
Dysentery (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 1 (1)
Haemophilus infection (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 2 (2)
Lower respiratory tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Malaria (Infections and infestations) | 1 (1) | 0 (0)
Mycoplasma infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 12 (12) | 6 (6)
Pneumonia bacterial (Infections and infestations) | 2 (2) | 3 (3)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2) | 1 (1)
Tuberculous pleurisy (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 2 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Burns first degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Electric shock (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 1 (1)
Heart rate irregular (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperosmolar hyperglycaemic state (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Astrocytoma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Cerebral haematoma (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrospinal fluid leakage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 3 (4)
Cerebrovascular disorder (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Monoparesis (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 3 (3) | 1 (1)
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Aggression (Psychiatric disorders) | 0 (0) | 1 (1)
Bipolar I disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Stress (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Pelvi-ureteric obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (1)
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Menometrorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 35 (38) | 36 (39)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Vocal cord disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
≥ 60 days prior to submission of material for publication/presentation, Institution and PI shall jointly provide AZ with material for review. No publication/presentation may include any of AZ's Confidential Information without AZ's written approval. AZ can request Inst. and PI to withhold material from submission for publication/presentation for an additional 90 days to allow AZ to establish and preserve its proprietary rights in the material being submitted for publication or presentation.